CLINICAL TRIAL: NCT00368394
Title: Dose-Exposure-Response Relationship of Insulin Glulisine (HMR1964) in Subjects With Type 1 Diabetes Mellitus Assessed With the Euglycemic Clamp Technique Using the Biostator (TM)
Brief Title: Dose-Exposure-Response in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HMR1964/1019; HMR1964
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-08

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Insulin glulisine; Euglycaemic clamp; Diabetes mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin glulisine

SUMMARY:
To investigate the dose-exposure-response relationship of insulin glulisine (HMR1964) after single subcutaneous injections of 0.075, 0.15 and 0.3 U/kg body weight with the euglycaemic clamp technique using the Biostator (TM).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-01

PRIMARY OUTCOMES:
Outcome measures: Glucose infusion rate, insulin concentrations.
Outcome:In T1DM, glulisine, like RHI, displays dose proportionality in exposure over the dose range 0.075 to 0.3 U/kg, which partly only translates into dose proportionality in glucodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Rave Dr, med, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Sanofi-Aventis, Neuss, Germany

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com